CLINICAL TRIAL: NCT04458207
Title: Cognitive Changes and Neural Correlates After Rehabilitation of Masticatory Function in Older Adults - an Intervention Study
Brief Title: Cognitive Changes and Neural Correlates After Rehabilitation of Masticatory Function in Elderly -an Intervention Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Folktandvården Stockholms län AB (Other Government)
Collaborators: Karolinska Institutet (Other); Eastmaninstitutet (Other)
Responsible Party: Principal Investigator, Linn Hedberg, DDS, Senior Consultat, PhDs, Folktandvården Stockholms län AB
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tugg&Tänk
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-03

CONDITIONS: Chewing Problem; Cognitive Decline; Magnetic Resonance Imaging; Degenerative; Dementia; Mastication Disorder; Neurocognitive Dysfunction
Keywords: Magnetic resonance imaging; Chewing efficiency; Cognitive impairment; Masticatory dysfunction; Prosthetic rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Cognition Disorders

STUDY DESIGN:
Intervention Model Description: Longitudinal randomized controlled trial. After screening and informed consent the participants are randomly allocated to exeperimental or control group. Both groups undergoing intervention but the participants in the control group undergo one more test before the intervention to rule out the test-retest effect.
Masking Description: The investigator doing the cognitve assements is not informed about the allocation of the participants.It is not possible to mask the participants during the neuropsycological assessements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (EG), the immediate rehabilitation group (Experimental): The experimental group will begin with the rehabilitation immediately after the first measurement of cognitive tests (pre-test). Three months after complete rehabilitation the first post-test (post-test 1) will be conducted on all participants. Participants will be recalled after about a year for a long-term follow up (post-test 2). The OHIP-14, chewing function test, saliva samples, neuropsychological assessments together with MRI assessments will also be recorded at different time points (i.e., pre-test, post-test 1 and post-test 2).
  Interventions: Procedure: Oral prosthetic rehabilitation
- Control group (CG), the test-retest group (Active Comparator): The control group will be tested with the cognitive tests two times (pre-test + post-test 1) at an interval of about three months or more inbetween tests and before the onset of the prosthodontic rehabilitation. Three months after complete rehabilitation the post-test (post-test 2) will be conducted on all participants. Further, participants will be recalled after about a year for a long-term follow up (post-test 3). The OHIP-14, chewing function test, saliva samples, neuropsychological assessments together with MRI assessments will also be recorded at these time points (i.e., pre-test, post-test 1, post-test 2 and post-test 3).
  Interventions: Procedure: Oral prosthetic rehabilitation

INTERVENTIONS:
Procedure: Oral prosthetic rehabilitation — Individual treatment options will be discussed with the participants individually and rehabilitation will be provided as agreed by the dentist and the participant. The rehabilitation will include fixed prosthodontics. The procedures will involve a control phase involving scaling, root planing oral hygiene instructions etc., extractions and bone augmentation when needed and temporary removable dentures. Restoration of the lost vertical dimension (if needed) with occlusal splints, tooth preparations, placement of dental implants (if needed) and finally cementation of dental crowns. The rehabilitation phase is estimated to take approximately 3-18 months, or more.

SUMMARY:
Today in elderly tooth loss and loss of oral function is widespread, but it is an underexplored modifiable risk factor potentially contributing to the development of dementia. In this interventional study a "cause-effect" relationship between mastication and cognition in humans will be investigated.

A total of eighty (80) participants, 65-80 years of age, indicated for prosthodontic rehabilitation will be randomly assigned to either the experimental or the control group. Participants will be randomized into two different groups, measurements are going to be conducted before and after prosthetic rehabilitation. The difference between the two groups is that the control group are going to do two measurements before undergoing the rehabilitation, this to control for the test-re-test effect.

The aim with this study is to determine if the rehabilitation of chewing function will cause changes in the neurocognitive assessments of episodic memory and learning.

DETAILED DESCRIPTION:
* Dementia is a general term of several neurodegenerative diseases that jointly affects approximately 7% of the general population older than 65 years, and 30% older than 80 years (O'Brien, 2003). Importantly, these statistics are expected to almost double every 20 years (Prince, 2013), making disorders of cognition a priority for healthcare (O'Brien, 2014).
* Animal and human studies have shown associations with mastication and cognitive function through the medial temporal lobe (i.e., hippocampus) and its role in learning and memory. (Ono, 2010. Weijenberg, 2011. Ohkubo, 2012. Teixeira, 2014. Klineberg, 2014)
* Although tooth loss and loss of oral function is widespread in older people, it is still an underexplored modifiable risk factor contributing to the development of dementia.
* The aim of this study is to conduct an intervention study on elderly people where rehabilitation of masticatory functions is performed and evaluated, with cognitive measures and brain imaging, to investigate a "cause-effect" relationship between mastication and cognition in humans.
* The hypothesis is that rehabilitation of masticatory function will improve cognition primarily in the performance of episodic memory and executive function tests along with the corresponding neural changes mainly in hippocampus and prefrontal cortex.
* A total of eighty (80) participants, 65-80 years of age, indicated for prosthodontic rehabilitation at Eastmaninstitutet (Stockholm, Sweden) will be randomly assigned to either the experimental or the control group. The difference between the groups is that the participants in the experimental group will begin with the rehabilitation immediately after the first measurement while the control group will do one more measurement before the onset of the rehabilitation procedure. The two measurements conducted before treatment in the control group are to rule out for test-retest effects. Three months and one year after completed prosthodontic treatment participants will conduct the last measurements, as a post-test to evaluate potential treatment effect.
* The neuropsychological assessments will be conducted together with MRI assessments, oral health-related quality of life instrument, chewing function test (two coloured chewing gum) and saliva samples recorded at different time points (i.e., pre-test, post-test 1, post-test 2, post-test 3) in both the groups.
* The data from the study will be entered in a Microsoft Excel sheet and exported to Statistics is a software package SPSS Inc, Statistica, StatSoft Inc (or similar advanced analytics software package for analysis). The result from the cognitive testing will be analysed as repeated measure Analysis of covariance (ANCOVAs) with groups (experimental and control) and time (pre- and post-rehabilitation) as factors. Group-by-time interaction, main effect of group, and main effect of time will be evaluated. To compare the magnitude of gains, the effect size (partial eta-square) will also be calculated. By using time-length between pre- and post-tests as a covariate of interest with aiming to better control group differences. Models that mainly predicts cognitive test measures (neuropsychological assessments) will by developed to predict the intervention outcomes. Predictive ability is defined as the amount of variance in the outcome that can be explained by pre-test cognitive status (slope method). Explained variance in outcome will be obtained by analysing linear regressions.
* Preprocessing and statistical analyses of MRI data will be performed with Statistical Parametric Mapping (SPM) run in Matlab (MathWorks). Movement correction will be performed by realign and unwarp to the first image in the series. To consider group-specific anatomical brain differences, all participants will be normalized to Monteral Neurological Institute (MNI) echoplanar-imaging template. Cortical thickness measures will not be normalized but rather used in their raw form. For cortical segmentation, a Freesurfer pipeline will be applied to the MRI images to produce regional cortical thickness and volumetric measures. To investigate rehabilitating-related changes repeated measures ANCOVAs will be performed with the groups (experimental and control) and time (pre- and post-rehabilitation) as factors. The Bonferroni-Holm method will be used to control for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* 65-80 years of age at start
* Impaired chewing ability (Eichner index B2-B4, C1-C4)
* Dental rehabilitation with fixed prosthodontics, implant and/or tooth supported (overdentures included) >10 occluding units
* Mini Mental State Examination (MMSE) score >25

Exclusion Criteria:

* Brain trauma or stroke <6 months
* Neurological disease (stroke, dementia, Alzheimer disease, Parkinson disease).
* Intellectual disability
* Psychological disorders
* Participants with chronic pain, depression or sleeping disorders
* Daily analgesic medication that may affect cognitive and/or executive performance of the brain
* Poor Swedish language skills, reading disabilities
* Severely reduced hearing or vision
* Prosthetic treatment with removable dentures (full or partial)

MRI exclusion criteria:

* Claustrophobia
* Difficulties in lying down in a supine position for about an hour, or any other difficulties related to the MRI head coil
* Participants with metal or medical implants in the body contraindicating MRI scan

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Visuospatial Memory Test Revised (BVMT-R) | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measuring non-verbal episodic memory. Measured in correct answers. Score: 0-36. A high score indicates a better performance.

SECONDARY OUTCOMES:
Change in Rey Auditory Verbal Learning Test (RAVLT). | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measuring verbal episodic memory. Measured in correct answers. Scale: 0-90. A high score indicates a better performance.
Change in Trail Making Test from Delis Kaplan Executive Function System (D-KEFS) | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measuring executive function. Measured in seconds and number of faults (maximum 150 seconds). A low score indicates a better performance.
Change in Digit-Span from Wechsler Adult Intelligence Scale (WAIS):IV | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measuring working memory. Measured in correct answers. Score: 0-48. A high score indicates better performance.
Change in Digit-symbol from Wechsler Adult Intelligence Scale (WAIS):IV | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measuring motor and mental speed. Measured in correct answers. Score: 0-135. A high score indicates better performance.
Change in Color-Word Interference Test from Delis Kaplan Executive Function System (D-KEFS word) | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measuring executive memory. Measured in seconds to complete test (maximum 90 seconds). Higher score indicates a poorer performance.
Change in verbal fluency from Delis Kaplan Executive Function System (D-KEFS-F) | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measuring executive memory. Measured in correct answer during a time limit (60 seconds). A high score indicates a better performance.
Title: Changes in blood perfusion in the brain tissue by measuring cerebral blood flow (CBF) in the brain over time with magnetic resonance imaging (MRI). | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measured with MRI using the Pseudo- Continuous Arterial Spin Labeling (pCASL) technique. The unit of measurement is ml of blood per 100 gram tissue per unit of time (ml/100g/min).
Changes in brain activity (BA) over time measured with magnetic resonance imaging (MRI). | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measuring changes in functional connectivity over time with MRI using the Blood Oxygen Level Dependent (BOLD) technique under resting state conditions.
Change of the masseter muscle volume (MMV) with magnetic resonance imaging (MRI). | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Measured with MRI using a PD-weighted SPACE sequence to determine the pre- and post-muscle volume. Volume increase indicates volume increase in muscle masseter.
Change in mixing ability (MA) two-coloured chewing gum (Orophys chewing gum) | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Two-coloured Orophys chewing gum. More mixed colour in the sample indicates better chewing ability.
Change in measure of cortisol level (CL) in saliva | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Biological measures. Low level of cortisol indicate lower stress hormone levels.
Change in Oral Health Impact Profile, short version (OHIP-14). | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Questionnaire measuring impact on daily life coast by oral problems. Scale: 0-56. Higher score indicates more impact or oral problems.
Change in psychological wellbeing the day of psychological assessment by using Hospital Anxiety and Depression scale (HAD). | 1: Baseline pre-test. 2: Change pre-test/post-test1, CG 3months after baseline, EG 3months after intervention (Int). 3: Change post-test1/post-test2, CG 3months after Int, EG 1year after Int. 4: Change post-test1/post-test2, CG 1year after Int.
  Questionnaire measuring Depression and Anxiety. Scale: 0-42. A low score indicate a more positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Trulsson, Prof. DDS, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Eastmaninstitutet Folktandvården Stockholm AB, Stockholm, Stockholm County
  - Eastmaninsitutet, Department of Prosthodontics, Stockholm

REFERENCES:
- [Background] O'Brien JT, Erkinjuntti T, Reisberg B, Roman G, Sawada T, Pantoni L, Bowler JV, Ballard C, DeCarli C, Gorelick PB, Rockwood K, Burns A, Gauthier S, DeKosky ST. Vascular cognitive impairment. Lancet Neurol. 2003 Feb;2(2):89-98. doi: 10.1016/s1474-4422(03)00305-3. PMID 12849265
- [Background] Prince M, Bryce R, Albanese E, Wimo A, Ribeiro W, Ferri CP. The global prevalence of dementia: a systematic review and metaanalysis. Alzheimers Dement. 2013 Jan;9(1):63-75.e2. doi: 10.1016/j.jalz.2012.11.007. PMID 23305823
- [Background] O'Brien JT, Markus HS. Vascular risk factors and Alzheimer's disease. BMC Med. 2014 Nov 11;12:218. doi: 10.1186/s12916-014-0218-y. PMID 25385509
- [Background] Ono Y, Yamamoto T, Kubo KY, Onozuka M. Occlusion and brain function: mastication as a prevention of cognitive dysfunction. J Oral Rehabil. 2010 Aug;37(8):624-40. doi: 10.1111/j.1365-2842.2010.02079.x. Epub 2010 Mar 2. PMID 20236235
- [Background] Weijenberg RA, Scherder EJ, Lobbezoo F. Mastication for the mind--the relationship between mastication and cognition in ageing and dementia. Neurosci Biobehav Rev. 2011 Jan;35(3):483-97. doi: 10.1016/j.neubiorev.2010.06.002. Epub 2010 Jun 12. PMID 20547177
- [Background] Ohkubo C, Morokuma M, Yoneyama Y, Matsuda R, Lee JS. Interactions between occlusion and human brain function activities. J Oral Rehabil. 2013 Feb;40(2):119-29. doi: 10.1111/j.1365-2842.2012.02316.x. Epub 2012 May 25. PMID 22624951
- [Background] Teixeira FB, Pereira Fernandes Lde M, Noronha PA, dos Santos MA, Gomes-Leal W, Ferraz Maia Cdo S, Lima RR. Masticatory deficiency as a risk factor for cognitive dysfunction. Int J Med Sci. 2014 Jan 10;11(2):209-14. doi: 10.7150/ijms.6801. eCollection 2014. PMID 24465167
- [Background] Klineberg I, Palla S, Trulsson M. Contemporary relevance of occlusion and mastication. Int J Prosthodont. 2014 Sep-Oct;27(5):411-2. doi: 10.11607/ijp.2014.5.e. No abstract available. PMID 25191880
- [Derived] Hedberg L, Ekman U, Nordin LE, Smedberg JI, Skott P, Seiger A, Sandborgh-Englund G, Westman E, Kumar A, Trulsson M. Cognitive changes and neural correlates after oral rehabilitation procedures in older adults: a protocol for an interventional study. BMC Oral Health. 2021 Jun 9;21(1):297. doi: 10.1186/s12903-021-01654-5. PMID 34107933